CLINICAL TRIAL: NCT04046302
Title: Effect of Self-Administered Vaginal Dinoprostone on Pain Perception During Copper Intrauterine Device Insertion in Parous Women: a Randomized Controlled Trial
Brief Title: Vaginal Dinoprostone Administration Prior to an Intrauterine Device Insertion in Multiparous Women.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dinoprostone IUD pain
Record Dates: First submitted 2019-08-04; First posted 2019-08-06 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: IUD Insertion
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dinoprostone (Experimental): 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) self-inserted by the patients 3 hours before the scheduled IUD insertion appointment.
  Interventions: Drug: Dinoprostone
- placebo (Placebo Comparator): one tablet of placebo self-inserted by the patients 3 hours before the scheduled IUD insertion appointment.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dinoprostone — 1 vaginal tablet of dinoprostone (3mg) (prostin® E2, Pharmacia & Upjohn, Puurs, Belgium) self-inserted by participants 3 hours before scheduled IUD insertion appointment.
  Arms: dinoprostone
Drug: placebo — one tablet of placebo self-inserted by participants 3 hours before scheduled IUD insertion appointment.
  Arms: placebo

SUMMARY:
To investigate whether vaginal dinoprostone administered before intrauterine device (IUD) insertion reduces failed insertions, insertion-related complications, and pain in multiparous women.

DETAILED DESCRIPTION:
Women may experience pain and technical difﬁculties may be encountered when insertion of an intrauterine device (IUD) is attempted through a narrow cervical canal.IUD insertion- related complications and side effects are more common among women who had never delivered vaginally. Pain can be perceived during all steps of IUD insertion including the application of the tenaculum to the cervical lip, sounding the uterus and advancing the IUD introducer through the cervical canal inside the uterine cavity

ELIGIBILITY:
Inclusion Criteria:

* multiparous women aged over 18 years of age requesting an IUD for contraception, had a negative pregnancy test.

Exclusion Criteria:

* currently pregnant or were pregnant within 6 weeks of study entry
* had a prior attempted or successful IUD insertion
* had a history of a cervical procedure such as cone biopsy, Loop electrosurgical excision procedure, or cryotherapy
* any World Health Organization Medical Eligibility Criteria category 3 or 4 precaution to an IUD
* active vaginitis or cervicitis
* undiagnosed abnormal uterine bleeding
* pelvic inﬂammatory disease within the last 3 months
* ﬁbroids or other uterine abnormalities distorting the uterine cavity
* contraindication or allergy to dinoprostone.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
the difference in the pain intensity scores between the study groups | 5 minutes
  the difference in the pain intensity scores between the study groups by visual analog scale score which ranges from zero to 10.where zero represents no pain and 10 represents the most worst pain

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine Cairo university, Giza, Egypt

REFERENCES:
- [Derived] Ashour AS, Nabil H, Yosif MF, Hussein M, Mageed A Allah AA, Mahmoud M, Abdou H, Kholaif K, Mohamed Kotb MM, El Sharkawy M, Abdelhakim AM, Ali AS, Nassar SA, Abbassy AH, Ghamry NK, Abdel-Latif AA, Taher A, El Mahy M. Effect of self-administered vaginal dinoprostone on pain perception during copper intrauterine device insertion in parous women: a randomized controlled trial. Fertil Steril. 2020 Oct;114(4):861-868. doi: 10.1016/j.fertnstert.2020.05.004. Epub 2020 Jul 28. PMID 32732105